CLINICAL TRIAL: NCT04604847
Title: Postoperative Painful Chronicization After Knee Replacement Surgery : Exploratory Study of BDNF's Kinetics
Acronym: KNEE BDNF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL19_0192
Record Dates: First submitted 2020-10-12; First posted 2020-10-27 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Total Knee Arthroplasty; Chronic Postoperative Pain
Keywords: Chronic Postoperative Pain; Brain Derived Neurotrophic Factor
MeSH Terms: conditions — Pain, Postoperative | interventions — Hematologic Tests

STUDY DESIGN:
Intervention Model Description: Prospective study to analyze perioperative blood samples in patient after knee replacement surgery. Patients will be included in the study at the pre-anesthetic consultation. Serum BDNF levels will be measured preoperatively, 48h postoperatively, 3 and 6 months after surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Total knee arthroplasty (Other): patient operated for a total knee arthroplasty
  Interventions: Diagnostic Test: blood test

INTERVENTIONS:
Diagnostic Test: blood test — blood test to explore BDNF level

SUMMARY:
Chronic pain is an extremely disabling disease. It is a major public health problem due to the lack of effective therapy.

Chronic postoperative pain (CPOP) is defined by a painful symptomatology in the operated area unrelated to previous pain, present for more than 3 months, and without any link to surgical complication.

The prevalence of chronicization of postoperative pain is 30% after total knee arthroplasty.

Identification of clinical, biological and psychological profiles are crucial to prevent CPOP.

A biologic factor, Brain Derived Neurotrophic Factor (BDNF) produced by a variety of cells is a key regulator of neuroplasticity. BDNF is increasingly studied in the mechanisms of cerebral sensitization and pain chronicization. The role of BDNF in pain of patients remains to be explored in a prospective study. The aim of this observational study is to compare the kinetics of BDNF after total knee arthroplasty in patients with and without CPOP.

Patients will be included in the study at the preanesthetic consultation. Serum BDNF levels will be measured preoperatively, 48h postoperatively, 3 and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Social security affiliation
* Adult patients
* Signed informed consent
* Score ASA (American Society of Anesthesiology) 1-3
* Total knee arthroplasty

Exclusion Criteria:

* Patient unable to exercise consent
* Pregnant women
* Vulnerable people
* Patients not included in the postoperative rehabilitation program
* Patients unable to complete the pain assessment questionnaires
* Chronic pain patients (other than knee arthrosis)
* Neuropathic pain patients (beforehand)
* Inflammatory diseases, progressive cancer, sepsis, immunosuppression known

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
BDNF level | preoperative to 6 months after surgery
  assessed by ELISA technique

SECONDARY OUTCOMES:
Pain level | preoperative to 6 months after surgery
  evaluated by Visual Analog Scale (VAS)
Neuropathic pain diagnostic | preoperative to 6 months after surgery
  evaluated by neuropathic pain diagnostic questionnaire (DN4)
Postoperative rehabilitation | preoperative to 6 months after surgery
  evaluated by the Brief Pain Questionary (BPI)
Health related quality of life | preoperative to 6 months after surgery
  evaluated by the SF-12 Health Survey
Anxiety and Depression | preoperative to 6 months after surgery
  evaluated by the Hospital Anxiety and Depression scale (HAD)
Pain level perception | preoperative to 6 months after surgery
  evaluated by the The pain Catastrophizing Scale
Assessment of functional capacities in knee arthritis | preoperative to 6 months after surgery
  evaluated by the Western Ontario and McMaster Universities Arthritis Index (WOMAC)
Oxidative stress marker | preoperative to 6 months after surgery
  8-iso-prostaglandin F2α level by biochemical labeling

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and critical care, Lapeyronie University Hospital, Montpellier, France